CLINICAL TRIAL: NCT03340285
Title: Randomized, Single-blind, Parallel-group, Placebo-controlled Study to Evaluate the Effect of a New Combination of Nutraceuticals (AkP06) Without Monacolin K on Plasma Lipids and Glucose
Brief Title: Effects of a New Combination of Nutraceuticals (AkP06) Without Monacolin K on Plasma Lipids and Glucose
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Bruno Trimarco, PROF OF CARDIOLOGY, Federico II University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AkP_6
Record Dates: First submitted 2017-11-08; First posted 2017-11-13 (Actual); Last update posted 2019-07-30 (Actual); Status verified 2019-07

CONDITIONS: Cardiovascular Risk Factor

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AkP06 (Experimental): first two weeks: Placebo + prescribed Diet then 4 weeks AkP06 two tablet/day before meals + Diet
  Interventions: Dietary Supplement: AkP06
- Placebo (Placebo Comparator): first two weeks: Placebo + prescribed Diet then 4 weeks Placebo two tablet/day before meals + Diet
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: AkP06 — first 2 weeks: Placebo + Diet then 4 weeks AkP06 two tablet/day before meals + Diet
  Arms: AkP06
Dietary Supplement: Placebo — first 2 weeks: Placebo + Diet then 4 weeks placebo two tablet/day before meals + Diet
  Arms: Placebo

SUMMARY:
The study is designed evaluate the effects of a new combination of nutraceuticals (AkP 06) without Monacolin K on lipid and glucose metabolism.

The study will analyze the impact of 4 weeks treatment with Akp06 or placebo, according to a randomized scheme, on metabolic parameters in dyslipidemic subjects that do not require or not tolerate a statin therapy. In particular, it will assess the ability of AkP 06 to reduce the plasma levels of LDL cholesterol, HbA1C, glicaemia and fasting insulin and to increase those of HDL cholesterol.

In addition, effects on serum transaminase and creatine phosphokinase (CPK) concentration will be evaluated.

DETAILED DESCRIPTION:
The experimental design involves the construction of a placebo-controlled, randomized, single-blind, parallel-groups.

Patients with mild hypercholesterolemia, of both sexes and aged between 18 and 75 years, will be recruited, from the beginning of the study and for the next 2 weeks at the outpatients Hypertension Clinic.

The subjects will be enrolled in the 50/50% male/female ratio ± 10% comparable for age, in order to obtain a proper comparison between groups with similar demographic characteristics or not statistically different.

The subjects, selected on the basis of inclusion and exclusion criteria, will be divided into two groups, to a computer based randomization scheme to receive one of two different treatments, two tablet/day before meals of the new nutraceutical AkP06 (Akademy Pharma) containing Morus Alba and without Monacolin K, vs. two tablet/day of placebo, always before meals. During the first two weeks both groups will follow the prescribed diet and assume placebo tablets. At the end, blood tests (traditional metabolic parameters, blood glucose, HbA1C, fasting insulin, transaminase levels, CPK) will be performed. During the next 4 weeks a group will assume AkP06 (Akademy Pharma) containing Morus Alba and without Monakolin K, the other will assume placebo and everyone will continue to follow the prescribed diet. At the end of this period blood tests will be repeated. Tablets of AkP06 and placebo will be provided by Akademy Pharma free of charge

ELIGIBILITY:
Inclusion Criteria:

* Total Cholesterol<300 mg/dL
* Total Cholesterol>200 mg/dL
* Cardiovascular Risk<20%

Exclusion Criteria:

* Pregnancy
* Documented intolerance to one or more components of AkP06
* Previous cardiovascular events
* Familiar severe dyslipidemia
* Familiar high cardiovascular risk Hepatic or muscular disorders Subjects receiving lipid-lowering drugs

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2018-03-31 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
Reduction of LDL-Cholesterol levels | 4 weeks

SECONDARY OUTCOMES:
Increasing of HDL-Cholesterol levels | 4 weeks
Reduction of HbA1c levels | 4 weeks
Reduction of fastin insuline levels | 4 weeks
No alteration of transaminase levels | 4 weeks
No alteration of CPK levels | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Trimarco, Professor, Principal Investigator — FEDERICO II UNIVERSITY - NAPLES
Locations (1):
- Raffaele Izzo, Naples, Italy

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code